CLINICAL TRIAL: NCT01351337
Title: Clinical Efficiency of Motor Pathway Mapping Using Diffusion Tensor Imaging Tractography and Intraoperative Subcortical Stimulation in Cerebral Glioma Surgery
Brief Title: Functional Monitoring for Motor Pathway in Brain Tumor Surgery Within Eloquent Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Collaborators: Shanghai Municipal Science and Technology Commission (Other Government)
Responsible Party: Principal Investigator, Jinsong Wu, professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 07QA14008; 07QA14008 (Other Grant/Funding Number: The govermment of Shanghai, China)
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Results first posted 2015-04-20 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Glioma, Motor Pathway
Keywords: Diffusion tensor imaging, Glioma, Intraoperative monitoring, Pyramidal tract, Subcortical; stimulation, Tractography
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intraoperative functional monitoring (Other): intraoperative functional monitoring
  Interventions: Procedure: diffusion tensor tractography neuronavigation and intraoperative subcortical stimulation

INTERVENTIONS:
Procedure: diffusion tensor tractography neuronavigation and intraoperative subcortical stimulation — All of the patients underwent tumor resection assisted with combined use of Diffusion tensor tractography-integrated functional neuronavigation and intraoperative subcortical stimulation

SUMMARY:
Resection of brain tumors in eloquent areas involves the risk of postoperative motor deficits. For brain tumors within or adjacent to the eloquent area, maximizing tumor resection while preserving motor function is crucially important.we used DTI-based tractography to visualize the spatial relationship between brain lesions and the nearby pyramidal tract(PT) in patients with malignant brain tumors and confirmed functional connections of the illustrated PT by direct electrical stimulation. We evaluated the reliability of DTI-based tractography for PT mapping using intraoperative subcortical stimulation ) and the usefulness of the combination of two techniques.

DETAILED DESCRIPTION:
Adverse effects caused by electrical stimulation during the operation were recorded. All subjects adopted early postoperative MRI examinations (within 3 days) to evaluate both the extent of tumor resection and the integrity of the PTs. Muscle strength was assessed preoperatively and postoperatively.The Karnofsky Performance Scale (KPS) was adopted for grading functional status at the 6-month evaluation. Further tumor progression interval and survival analysis was conducted for each subject with high-grade glioma (HGG)

ELIGIBILITY:
Inclusion Criteria:

* patients with an initial imaging diagnosis of single, unilateral, supratentorial primary glioma (or intrinsic neoplasm).
* The lesions were involved in PTs, comprising cortical regions in the motor or somatosensory areas, cortical regions adjacent to the central gyrus, subcortical regions with an infiltrative progression along the PTs, and temporal or insular regions in relation to the internal capsule.
* MRI enabled preoperative identification of patients in whom maximal tumor resection was likely to be achieved, and close PT approach within resection cavity at the time of surgery was possible.

Exclusion Criteria:

* patients with secondary or recurrent gliomas (or intrinsic neoplasm), patients with contraindications for MRI or direct electrical stimulation, and patients in whom initial muscle strength grades of the affected extremities was 2/5 or lower.

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liangfu Zhou, Doctorate, Study Chair — Huashan Hospital
Locations (1):
- Hushan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Zhu FP, Wu JS, Song YY, Yao CJ, Zhuang DX, Xu G, Tang WJ, Qin ZY, Mao Y, Zhou LF. Clinical application of motor pathway mapping using diffusion tensor imaging tractography and intraoperative direct subcortical stimulation in cerebral glioma surgery: a prospective cohort study. Neurosurgery. 2012 Dec;71(6):1170-83; discussion 1183-4. doi: 10.1227/NEU.0b013e318271bc61. PMID 22986591

RESULTS

PARTICIPANT FLOW:
Groups:
- Intraoperative Functional Monitoring: intraoperative functional monitoring and diffusion tensor tractography
  All of the patients underwent tumor resection assisted with combined use of Diffusion tensor tractography-integrated functional neuronavigation and intraoperative subcortical stimulation
Period: Overall Study
Arm/Group | Intraoperative Functional Monitoring
Started | 58
Completed | 58
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Age (range), y 44 (10-72) Female/male, n/n 21/37
Arm/Group | Intraoperative Functional Monitoring
Number analyzed (Participants) | 58
Age, Continuous [Mean (Full Range); unit: years]
  Patients enrolled | 44 [10 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 37
Study Specific Measure [Tumor Location] [Number; unit: participants]
  Frontal lobe | 22
  Parietal lobe | 13
  Insular lobe | 12
  Temporal lobe | 11

OUTCOME MEASURES:

1. Primary Outcome: Extent of Tumor Resection
Description: Volumetric analysis was performed both before and after surgery by calculating the tumor volume on the images of enhanced 3-D MP-RAGE sequence for high-grade gliomas and FLAIR sequence for low-grade gliomas. The extent of tumor resection was the ratio of pre-op tumor volume over post-op tumor volume. Gross total resection refers to a 100% resection of the tumor volume; near-total resection refers to 95% to 100% resection; subtotal resection refers to 90% to 95% resection; partial resection refers to 75% to 90% resection; and biopsy refers to ,75% resection of the tumor volume for histological diagnosis.
Time Frame: within 3 days
Measure: Number; unit: participants
Arm/Group | Intraoperative Functional Monitoring
Number analyzed (Participants) | 58
participants
  gross total resection | 40
  near-total resection | 7
  subtotal resection | 7
  partial resection | 4

2. Secondary Outcome: Postoperative Motor Function and Long-time Functional Status
Description: Motor function was assessed early postoperatively (within 72 hours after the operation), and 1 month after discharge. The muscle strength of each subject was graded for both the upper and lower extremities with the Medical Research Council Scale. Grade 5: Muscle contracts against full resistance; Grade 4: Strength reduced, but contraction can still move joint against resistance; Grade 3: Strength further reduced such that joint can be moved only against gravity with examiner's resistance completely removed. Grade 2: Muscle can onlly move if resistance of gravity is removed. Grade 1: Only a trace or flicker of movement is seen or felt, or fasciculations are observed; Grade 0:No movement.
Time Frame: 3 days to 6 months after surgery
Measure: Number; unit: participants
Arm/Group | Intraoperative Functional Monitoring
Number analyzed (Participants) | 58
participants
  Normal | 41
  Short-term motor deficit | 11
  Long-term motor deficit | 6

3. Other Pre Specified Outcome: The Specificity, Sentitivity of DTI Tractography and Accordance Rate of DTI With DsCS Results
Description: The sensitivity of DTI tractography for PT mapping was calculated as the ratio between the number of subjects with positive DsCS results in the positive DTI zone (true positive) and the total number of subjects with positive DsCS results (true positive plus false negative). The specificity was measured as the ratio between the number of subjects with negative DsCS results in the negative DTI zone (true negative) and the total number of subjects with negative DsCS results (true negative plus false positive). The accordance rate of DsCS and DTI was measured as the ratio between the number of subjects with either a true-positive or true-negative DsCS result and the total number of subjects.
Time Frame: During the operation
Measure: Number; unit: percentage of stimulation sites
Arm/Group | Intraoperative Functional Monitoring
Number analyzed (Participants) | 58
percentage of stimulation sites
  Sentitivity | 92.6
  Specificity | 93.2
  Accordance rate | 92.9

ADVERSE EVENTS:
Time Frame: Within1 week
Description: We recorded the peri-operative adverse events which might influence the postoperative motor function of each subject, including cavity bleeding, death.
Arm/Group | Intraoperative Functional Monitoring
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 0/58

LIMITATIONS AND CAVEATS:
The imaged motor pathway was reconstructed based on pre-opimages. An additional study that integrates real-time DTI tractography with high-field intraoperative MRI and DsCS for eloquent cerebral glioma surgery is currently underway in our department.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No